CLINICAL TRIAL: NCT05964699
Title: The Use of a Non-Incised Minimally Invasive Flap Procedure in Conjunction With Emdogain® MI Compared to Traditional SRCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2022-1175-CD-DCR
Record Dates: First submitted 2023-06-26; First posted 2023-07-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Periodontitis; Attachment Loss, Periodontal
MeSH Terms: conditions — Periodontitis; Periodontal Attachment Loss

STUDY DESIGN:
Intervention Model Description: Split mouth study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and outcome assessors are unaware of the assigned interventions. The care provider will know at this time of procedure what site will receive the intervention and what site will be the control site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Periodontal regeneration (Experimental): Regeneration will be attempted during root scaling and planing with the application of Emdogain and the use of a Videoscope.
  Interventions: Procedure: Minimally invasive periodontal therapy with use of Emdogain
- Control (Placebo Comparator): The control group will receive standard-of-care root scaling and planing without the application of Emdogain and the use of a Videoscope.
  Interventions: Procedure: Minimally invasive periodontal therapy without the use of Emdogain

INTERVENTIONS:
Procedure: Minimally invasive periodontal therapy with use of Emdogain — Scaling of root with assisted use of the Videoscope and regrowth of attachment by the use of Emdogain.
  Arms: Periodontal regeneration
Procedure: Minimally invasive periodontal therapy without the use of Emdogain — Scaling of root with assisted use of the Videoscope.
  Arms: Control

SUMMARY:
This study is designed to evaluate the use of Emdogain® MI in a procedure where a significant portion of the lining of the sulcus is removed by curettage (similar to the traditional clinical procedure described as "gingival curettage") to the point of tissue mobility. This will be designated as a "non-incised minimally invasive flap access procedure". A videoscope will be utilized to assist with the requirement to adequately visualize and debride the root surface. This research project will define the approach used as a "non-incised minimally invasive flap access" approach and will be a modification of recognized minimally invasive techniques. This modification will be made by Dr. Harrel who first describe the minimally invasive periodontal approach and defined minimally invasive periodontal procedures in 1995.

DETAILED DESCRIPTION:
The use of a non-incised minimally invasive flap procedure in conjunction with Emdogain MI compared to traditional scaling and root planing.

Background

The product Emdogain® MI is designed for use in a minimally invasive approach to periodontal treatment. This product is being marketed for what is termed a "flapless" procedure whereby scaling and root planing (SRP) is performed, the root surface is "visualized", debrided, and conditioned with EDTA (PrefGel), and then Emdogain® MI is inserted between the root surface and the sulcus tissue to reduce inflammation and stimulate reattachment.

The approach described above has met with mixed success. The concerns are associated with difficulty in the visualization of the sulcus and the difficulty in removing root accretions (calculus) with the "flapless" approach.

Purpose

This study is designed to evaluate the use of Emdogain® MI in a procedure where a significant portion of the lining of the sulcus is removed by curettage (similar to the traditional clinical procedure described as "gingival curettage") to the point of tissue mobility. This will be designated as a "non-incised minimally invasive flap access procedure". A videoscope will be utilized to assist with the requirement to adequately visualize and debride the root surface. This research project will define the approach used as a "non-incised minimally invasive flap access" approach and will be a modification of recognized minimally invasive techniques. This modification will be made by Dr. Harrel who first describe the minimally invasive periodontal approach and defined minimally invasive periodontal procedures in 1995. Note: No portion of this research will be utilized for a new or modified FDA application.

This study is being performed to assess if the use of Emdogain® MI in conjunction with SRP and videoscope visualization can provide better treatment outcomes, resulting in the improvement of periodontal clinical parameters when compared to traditional SRP and videoscope visualization without the use of Emdogain® MI.

Rational of the study

Hypothesis - To demonstrate that Emdogain® MI applied to an adequately visualized and debrided root surface using a non-incised minimally invasive flap access procedure will result in improvement of periodontal clinical parameters when compared to traditional SRP without the use of Emdogain® MI.

Primary End Point

Report the amount of improvement in clinical markers (PD, CAL, recession/keratinized tissue, BOP, PI) following non-incised minimally invasive flap periodontal procedures performed with direct videoscope visualization and root debridement followed by the application of Emdogain® MI compared to SRP without the use of Emdogain® MI.

Secondary End Points

Report the time necessary to perform the test procedures, compare the patient perception of the test and control procedures such as immediate post-treatment discomfort and impact on life activities, and report the patient perception of long-term post-treatment function and esthetics.

Indication

The non-incised minimally invasive flap procedure is indicated for isolated defects on teeth located in esthetic areas that initially present with moderate pocket depth and minimal radiographic detectable bone loss. In routine/traditional clinical practice, these isolated more advanced defects will often be treated by non-surgical/non-regenerative procedures i.e. scaling and root planing, only. The use of SRP only will frequently result in less than a complete resolution of the periodontal defect. The proposed non-incised minimally invasive flap procedure will be indicated and performed as an adjunct for isolated deeper pockets encountered during routine quadrant SRP.

Materials and Methods

This will be a single masked clinical outcomes study. Ethical approval will be obtained from the Texas A&M University IRB and study ethical standards and registration will follow the IRB's established guidelines.

Patients will be selected from patients presenting for routine periodontal treatment at Texas A&M University College of Dentistry department of Periodontology. Prior to entering the study, patients will have radiographs and periodontal charting performed. Based on the pre-study evaluation and radiographs, patients will be treatment planned for non-surgical (SCRP) periodontal treatment as initial therapy. A review of the initial records will determine potential candidates for this study. The study teeth will be limited to bicuspid and cuspid teeth. To be included in the study, patients will present with generalized periodontitis with isolated pockets depths of 5 to <7 mm on bicuspid and cuspid teeth, no more than 1 mm of radiographic bone loss apparent on study teeth, and at least 2 mm of attachment loss. To qualify for the study there will need to be two similar teeth in a single patient meeting the criteria for isolated pockets in two separate quadrants. One site will be randomly assigned as a test site (non-incised minimally invasive flap procedure with Emdogain® MI) and the other will be assigned as the control site (SRP and Videoscope only).

Test and control site breakdown:

* Standard deep cleaning (SRP) on all teeth in one quadrant and the use of a small camera (Videoscope) on one tooth on that side (control tooth).
* On the other quadrant you will receive a standard deep cleaning (SRP) of all teeth in that quadrant and the use of a small camera called a videoscope and the protein gel which is what we call the closed access procedure on one tooth (research / test tooth).

Inclusion criteria will be patients between 30 and 75 years of age, in general good health (ASA I or II), smoke less than 10 cigarettes or equivalent per day, have no antibiotics for the past 90 days, and not taking medications that are known to inhibit or slow healing. Exclusion criteria will be pregnant or lactating patients, active periodontal treatment in the last 6 months, smokers of greater than 10 cigarettes per day, and patients with serious medical conditions.

On the day of treatment, a calibrated blinded evaluator will record all clinical parameters for the test and control teeth. These will include oral hygiene level, BOP, PD, CAL, keratinized gingival width, and standardized photographs. Radiographs will be taken of the test and control sites. All patients will be administered adequate local anesthetic for pain control in the areas to be treated. The operator will not be informed at this point as to the control and test teeth. All sites will have SRP performed utilizing the videoscope for intersulcular root visualization. The endpoint of SCRP will be when the therapist can not see or feel any calculus (tartar) or roughness on the root surface. Within the routine clinical limits of SCRP, the sulcus may be curetted and the soft tissue removed to the point that the clinician feels there is adequate access for evaluation and debridement of the root surface. At that point, the designated oral sites will be revealed to the treating therapist as having been designated to test or control by random assignment.

No further treatment will be performed on the control site with the exception of placing saline solution in the control site in a manner mimicking the use of Emdogain® MI in the test site. In the test sites, the sulcus will be curetted to the point that the tissue surrounding the teeth becomes moveable with gentle finger pressure. The curettage will be performed using routine periodontal curettes designed for sulcular curettage. No incisions will be made. When the tissue is moveable, the test site will be described as having non-incised minimally invasive flap access. The "flap" designation will be made because the tissue is moveable as is the case with traditional "flap" procedures. Further visualization of the root surface will be performed using the videoscope and, as necessary, the root on the test and control tooth will be further debrided of all remaining visible calculus and roughness. It will be recorded if there is or is not further material to be removed i.e. if there is material remaining after routine SCRP. Neutral EDTA (PrefGel) will be used to condition the root surface and Emdogain® MI applied to the test tooth following the manufacturers' instructions. In both control and test sites, the tissue will only be stabilized post-treatment by applying finger pressure. No sutures will be used. The time necessary to complete the additional procedures (beyond SCRP) on the test tooth will be recorded.

Patients will be seen for postoperative evaluation at one week, 3 months, and 6 months. The dental cleanings (gum maintenances / periodontal maintenance) and follow-up visits are part of standard of care and are not for research-only purposes. Patients who undergo deep cleaning should have their maintenance appointments (gum maintenances) every 3 months as part of standard of care.

Oral hygiene will be reinforced and photographs made at the one-week visit but no clinical measurements will be made. Clinical parameters will be measured and recorded by a calibrated blinded evaluator at the 3 and 6-month evaluation followed by a routine periodontal maintenance procedure. A radiograph using paralleling technique will be obtained prior to treatment and at the 6-month postsurgical evaluation. All patients will be asked to fill out a VAS pain scale for the test and control areas the evening following the procedure and at each post-surgical evaluation appointment.

ELIGIBILITY:
Inclusion Criteria:

To participate in this study, you must present:

* Generalized gum disease with isolated pocket depths of 5 mm to less than 7 mm on bicuspid and cuspid teeth.
* At least 2 mm of attachment loss.
* Need to have two similar teeth meeting the criteria for isolated pockets on two other quadrants of the mouth.
* Need to be between 30 and 75 years of age.
* Be in good health.
* Smoke less than 10 cigarettes or equivalent per day.
* No antibiotics for the past 90 days.
* Not be taking medications that are known to inhibit or slow healing.

Exclusion Criteria:

You are not eligible if:

* You are pregnant.
* You are breast feeding.
* Received gum treatment in the last 6 months.
* Smoke more than ten cigarettes per day.
* You have any serious medical conditions.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Attachment level change. | The attachment change will be determined from baseline to the 3 month follow-up and at the 6-month follow-up examination.
  Attachment change will be determined by measuring clinical probing depth and gingival marginal level with an UNC probe. The clinical attachment level is the distance from the cemento-enamel junction to the tip of a periodontal probe during periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement.
Probing depth change. | Probing depth change will be determined from baseline to the 3 month follow-up and 6 month follow-up.
  Probing depth change will be determined with an UNC probe during clinical examination on the control and test sites. Probing depth will be recorded on the periodontal examination chart at the initial visit, the 3-month and 6-month follow-up appointments. Probing depth is the distance from the soft tissue (gingiva or alveolar mucosa) margin to the tip of the periodontal probe.
Gingival margin level / recession change. | Gingival margin level / recession level change will be determined from baseline to the 3 month follow-up and 6 month follow-up.
  Gingival margin level / recession will be determined with an UNC probe during clinical examination on the control and test sites. Gingival margin level / recession will be recorded on the periodontal examination chart at the initial visit, the 3-month and 6-month follow-up appointments. The migration of the marginal soft tissue to a point apical to the cemento-enamel junction of a tooth or the platform of a dental implant is defined as recession.
Bleeding on probing change. | The bleeding of probing change will be determined from the baseline to the 3 month follow-up and 6 month follow-up.
  Bleeding on probing will be determined with an UNC probe during clinical examination on the control and test sites. Bleeding of probing sites will be recorded on the periodontal examination chart at the initial visit, the 3-month and 6-month follow-up appointments. Bleeding on probing happens when induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth.
Biofilm presence change. | Biofilm presence change will be determined from the baseline to the 3 month follow-up and 6 month follow-up.
  Biofilm presence will be determined with an UNC probe during clinical examination on the control and test sites. Biofilm will be recorded on the periodontal examination chart at the initial visit, the 3-month and 6-month follow-up appointments. Dental plaque is the prototypical example of a biofilm.

SECONDARY OUTCOMES:
Time necessary to perform the test procedures | 1 day (Time necessary to perform the test procedure at the initial appointment.)
  Report the time necessary to perform the test procedures - non-incised minimally invasive flap procedure in conjunction with Emdogain.
VAS pain scale 24 hours after appointment. | 24 hour follow-up.
  VAS pain scale for the test and control areas the following the procedure at 24 hours after appointment. The VAS scale is a tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.
VAS pain scale 1 week after appointment. | 1 week following the procedure.
  VAS pain scale for the test and control areas 1 week following the procedure. The VAS scale is a tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M School of Dentistry, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No